CLINICAL TRIAL: NCT03478514
Title: A Phase II Study of Palbociclib (PD-0332991) in Combination With Ibrutinib in Patients With Previously Treated Mantle Cell Lymphoma
Brief Title: Phase II Palbociclib +Ibrutinib in Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFT-32
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma; B Cell Lymphoma
Keywords: mantle cell lymphoma; B-cell lymphoma; palbociclib
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, B-Cell | interventions — palbociclib; ibrutinib

STUDY DESIGN:
Intervention Model Description: The proposed study is a single-arm, multi-center, open-label phase II study of the combination of palbociclib and ibrutinib in patients with previously treated mantle cell lymphoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients will receive palbociclib at 100 mg oral once a day for 21 days, followed by 7 days off.
  Ibrutinib will be administered at 560 mg oral continuously.
  Interventions: Drug: Palbociclib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Palbociclib — Taken at 100 mg once daily for 21 days, followed by 7 days off
  Other Names: Ibrance; PD-0332991
Drug: Ibrutinib — 560 mg taken orally all patients throughout the study
  Other Names: Imbruvica

SUMMARY:
The proposed study is a single-arm, multi-center, open-label phase II study of the combination of palbociclib and ibrutinib in patients with previously treated mantle cell lymphoma to evaluate the efficacy of this combination, with the primary objective of the study being to assess median PFS and the secondary objectives to include ORR, CR, DOR, OS and toxicity. Subjects will be enrolled and treated with palbociclib and ibrutinib with each cycle of therapy being 28 days. Treatment will be based on the recommended phase II dose (RP2D) from the phase I combination trial.

DETAILED DESCRIPTION:
Treatment will consist of:

* Palbociclib administered at 100 mg oral once daily for 21 days on followed by 7 days off
* Ibrutinib administered at 560 mg oral continuously

Patients will continue to receive study drugs until disease progression, unacceptable toxicity, or withdrawal of consent. If at any time one of the agents is held due to toxicity, the other agent may be continued in those patients who are receiving clinical benefit.

Response will be assessed by PET/CT and/or CT every 3 cycles while on therapy for the first year and then every 6 cycles thereafter until disease progression or at the investigator's discretion if otherwise medically indicated. A PET will be required to confirm CR. A bone marrow biopsy will be performed in patients with bone marrow involvement at the start of therapy to confirm complete response once patients have otherwise met criteria for CR.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed MCL as defined by the World Health Organization. All patients must have either t(11;14) by karyotype or fluorescent in-situ hybridization (FISH) or positive immunohistochemistry (IHC) for cyclin D1.
2. Subjects must have measurable disease defined as at least one tumor lesion of at least 1.5 cm by CT or MRI, PET positive lesion(s) or a peripheral blood CD5+, CD19+ lymphocyte count of at least 5,000 cells/µL.
3. Subjects must have received at least one prior systemic therapy.
4. Subjects who have received prior autologous stem cell transplant are eligible. Patients that have undergone prior allogeneic stem cell transplant will only be eligible if the patient is no longer taking immunosuppressive therapy and there are no significant ongoing transplant-related adverse effects.
5. Subjects must be age ≥ 18 years
6. ECOG performance status ≤ 2
7. Patients must have normal organ and marrow function as defined below:
8. Laboratory Values:

   * ANC ≥ 1000 cells/μL, unless bone marrow involvement in MCL, then ANC >500 cells/μL;
   * Platelets ≥ 75,000 cells/μL, unless bone marrow involvement in MCL, then platelets >30,000 cells/μL;
   * Calculated creatinine clearance ≥30mL/min;
   * AST or ALT ≤ 2.5x ULN;
   * Total bilirubin ≤ 1.5x ULN;
   * QTc ≤ 480 ms
9. Subjects must be able to provide written, informed consent
10. Subjects must have recovered from adverse events to ≤ grade 1 from prior therapies
11. Subjects must be able and willing to swallow and retain oral medication without a condition that would interfere with enteric absorption
12. Subjects may be receiving prednisone at a maximum dose of 20 mg orally daily for symptom control.
13. Serum or urine pregnancy test must be negative within 7 days of starting study treatment in women of childbearing potential. Women of childbearing potential and men with female partners who are able to become pregnant are required to use a highly effective form of barrier contraception for the duration of the study and for 90 days after the last dose of study drug. Adequate contraception is defined as abstinence or two forms non hormonal contraception, which is a combination of two forms of the following:

    * Condom with spermicidal foam/gel/cream/suppository
    * occlusive cap (diaphragm or cervical vault caps) with spermicidal
    * non hormonal intrauterine device (IVD)
14. No evidence of active hepatitis B or C infections (i.e., no positive serology for anti-HBc or anti-HCV antibodies)
15. HBV seropositive patients (HBsAg +) are eligible if they are closely monitored for evidence of active HBV infection by HBV DNA testing and receive suppressive therapy with lamivudine or other HBV suppressive therapy until 6 months after the last rituximab dose.
16. Patients with HIV infection are eligible, provided they meet the following:

    * No evidence of coinfection with hepatitis B or C
    * CD4+ cell count ≥ 400/mm3
    * No evidence of resistant strains of HIV
    * If not on anti-HIV therapy, HIV viral load < 10,000 copies HIV RNA/mL If on anti-HIV therapy, HIV viral load < 50 copies HIV RNA/mL
    * No history of AIDS-defining conditions
    * No use of strong CYP3A4/5 inhibitors or inducers

Exclusion Criteria:

1. Subjects that have received prior CDK4/6 inhibitor will not be eligible.
2. Subjects that have received any prior BTK inhibitor > 90 days prior to enrollment will not be eligible.
3. Subjects with known or suspected CNS involvement.
4. Concurrent therapy with other investigational products.
5. History of allergic reactions attributed to compounds of chemical or biologic composition similar to palbociclib.
6. Subjects receiving any medications or substances that are strong or moderate inhibitors or strong inducers of CYP3A isoenzymes within 7 days of starting study treatment (See Appendix II).
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Subjects with myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities are not eligible. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
9. Pregnant women, or women of childbearing potential without a negative pregnancy test (serum or urine) within 7 days prior to registration, irrespective of the method of contraception used, are excluded from this study because the effect of palbociclib on a developing fetus is unknown. Breastfeeding should be discontinued prior to study entry.
10. Subjects must agree to use barrier contraceptive methods throughout the study period up until at least 90 days post last palbociclib dose.
11. Subjects with clinically significant history of liver disease, including viral or other known hepatitis, current alcohol abuse, or cirrhosis, etc.
12. Subjects with another active malignancy that limits survival.
13. Subjects with a bleeding diathesis are not eligible.
14. Subjects with transfusion-dependent thrombocytopenia are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 42 months
  Time interval between registration and progression or death

SECONDARY OUTCOMES:
Overall survival | 42 months
  time from registration to death due to any cause
Duration of response | 42 months
  Time from documentation of tumor response to disease progression
Overall Response Rate | 42 Months
  Proportion of patients with reduction in tumor burden of a predefined amount
Complete Response | 42 Months
  Disappearance of all non-target lesions and normalization of tumor marker level
Toxicity: Incidence and severity of adverse events by summaries of toxicity data/contingency tables | 42 Months
  Evaluation of incidence and severity of adverse events by summaries of toxicity data/contingency tables

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Kami Maddocks, MD, Study Chair — Ohio State University
Locations (9):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Joseph Mercy Hospital Cancer Care Center, Ypsilanti, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina - Hollings Cancer Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herrmann A, Hoster E, Zwingers T, Brittinger G, Engelhard M, Meusers P, Reiser M, Forstpointner R, Metzner B, Peter N, Wormann B, Trumper L, Pfreundschuh M, Einsele H, Hiddemann W, Unterhalt M, Dreyling M. Improvement of overall survival in advanced stage mantle cell lymphoma. J Clin Oncol. 2009 Feb 1;27(4):511-8. doi: 10.1200/JCO.2008.16.8435. Epub 2008 Dec 15. PMID 19075279
- [Background] Medema RH, Herrera RE, Lam F, Weinberg RA. Growth suppression by p16ink4 requires functional retinoblastoma protein. Proc Natl Acad Sci U S A. 1995 Jul 3;92(14):6289-93. doi: 10.1073/pnas.92.14.6289. PMID 7603984
- [Background] Fry DW, Bedford DC, Harvey PH, Fritsch A, Keller PR, Wu Z, Dobrusin E, Leopold WR, Fattaey A, Garrett MD. Cell cycle and biochemical effects of PD 0183812. A potent inhibitor of the cyclin D-dependent kinases CDK4 and CDK6. J Biol Chem. 2001 May 18;276(20):16617-23. doi: 10.1074/jbc.M008867200. Epub 2001 Feb 6. PMID 11278443
- [Background] Marzec M, Kasprzycka M, Lai R, Gladden AB, Wlodarski P, Tomczak E, Nowell P, Deprimo SE, Sadis S, Eck S, Schuster SJ, Diehl JA, Wasik MA. Mantle cell lymphoma cells express predominantly cyclin D1a isoform and are highly sensitive to selective inhibition of CDK4 kinase activity. Blood. 2006 Sep 1;108(5):1744-50. doi: 10.1182/blood-2006-04-016634. Epub 2006 May 11. PMID 16690963
- [Background] Wang ML, Rule S, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Li L, Zhang L, Newberry K, Ou Z, Cheng N, Fang B, McGreivy J, Clow F, Buggy JJ, Chang BY, Beaupre DM, Kunkel LA, Blum KA. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med. 2013 Aug 8;369(6):507-16. doi: 10.1056/NEJMoa1306220. Epub 2013 Jun 19. PMID 23782157
- [Background] Martin P, Bartlett NL, Blum KA, Park S, Maddocks K, Ruan J, Ridling L, Dittus C, Chen Z, Huang X, Inghirami G, DiLiberto M, Chen-Kiang S, Leonard JP. A phase 1 trial of ibrutinib plus palbociclib in previously treated mantle cell lymphoma. Blood. 2019 Mar 14;133(11):1201-1204. doi: 10.1182/blood-2018-11-886457. Epub 2019 Jan 28. PMID 30692121
- [Background] Chiron D, Di Liberto M, Martin P, Huang X, Sharman J, Blecua P, Mathew S, Vijay P, Eng K, Ali S, Johnson A, Chang B, Ely S, Elemento O, Mason CE, Leonard JP, Chen-Kiang S. Cell-cycle reprogramming for PI3K inhibition overrides a relapse-specific C481S BTK mutation revealed by longitudinal functional genomics in mantle cell lymphoma. Cancer Discov. 2014 Sep;4(9):1022-35. doi: 10.1158/2159-8290.CD-14-0098. Epub 2014 Jul 31. PMID 25082755
- [Background] Leonard JP, LaCasce AS, Smith MR, Noy A, Chirieac LR, Rodig SJ, Yu JQ, Vallabhajosula S, Schoder H, English P, Neuberg DS, Martin P, Millenson MM, Ely SA, Courtney R, Shaik N, Wilner KD, Randolph S, Van den Abbeele AD, Chen-Kiang SY, Yap JT, Shapiro GI. Selective CDK4/6 inhibition with tumor responses by PD0332991 in patients with mantle cell lymphoma. Blood. 2012 May 17;119(20):4597-607. doi: 10.1182/blood-2011-10-388298. Epub 2012 Mar 1. PMID 22383795